CLINICAL TRIAL: NCT03313531
Title: Calibrated Automated Thrombogram: A Scandinavian Multicenter Study
Brief Title: Evaluation of a Standardized Protocol for Thrombin Generation Assay
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Other Study IDs: TGA1
Record Dates: First submitted 2017-10-12; First posted 2017-10-18 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-01

CONDITIONS: Hemophilia A
Keywords: Thrombin generation; variability; level of agreement; hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Study group 1: Patients with severe hemophilia A
  Interventions: Diagnostic Test: Thrombin Generation Assay
- Study group 2: Healthy volunteers
  Interventions: Diagnostic Test: Thrombin Generation Assay
- Study group 3: Healthy volunteers ) that at previous measurements have been shown to have a TGC>2SD of the median of the control population.
  Interventions: Diagnostic Test: Thrombin Generation Assay
- Treated HA person: One patient with severe hemophilia A (HA) will be treated with two factor FVIII concentrates, one with standard half- life (Advate™) and one with a pro-longed half-life (Adynovate™) at two separate occasions
  Interventions: Diagnostic Test: Thrombin Generation Assay; Drug: Treatment with recombinant coagulation factor

INTERVENTIONS:
Diagnostic Test: Thrombin Generation Assay — Inter lab variation and level of agreement will be determined
Drug: Treatment with recombinant coagulation factor — To obtain a wide range of thrombingeneration levels, one person (Treated HA person) will recieve one injection of Advate and one injection of Adynovate respectively
  Groups: Treated HA person

SUMMARY:
This study is aims at determining the inter laboratory variation when using the thrombin generation assay calibrated automated thrombogram (TGA CAT). It is thus, not a clinical trial in its usual meaning. However, to achieve relevant test samples one patient will be treated with two different study drugs as part of the trial and therefore, approval by Läkemedelsverket is needed. Test plasma samples will be sent out to five participating centers in the Scandinavian countries (Gothenburg and Stockholm, Sweden, Århus Denmark, Oslo Norway and Helsinki Finland) and coefficients of variance (CV) and level of agreement will be analyzed. To obtain representative plasma samples with a wide range of thrombin generation capacity (TGC), blood samples will be collected from research persons that has given informed consent to participate in the study. To obtain plasma with low TGC, blood samples will be drawn from patients with severe hemophilia (n=4)(study group 1), to obtain plasma with normal TGC, blood samples will be drawn from healthy volunteers (n=3)(study group 2) and to obtain plasma with high TGC, plasma will be collected from healthy volunteers (n=3)(study group 3) that at previous measurements have been shown to have a TGC>2SD of the median of the control population. Moreover, one patient with severe hemophilia A (HA) will be treated with two factor FVIII concentrates, one with standard half- life (Advate™) and one with a pro-longed half-life (Adynovate™) at two separate occasions (Treated HA person). By taking repeated blood samples after administration, samples with a wide range of FVIII levels and TGC:s will be obtained. Moreover, the effect of using plasmas with low, normal and high TGC for normalization will be investigated. Plasma samples will be collected as soon as approval from the Swedish medical agency (SMA) has been obtained, we count on sending them to participating centers March 2017. All laboratory measurements, data analysis and report writing will be concluded before December 31 2017.

DETAILED DESCRIPTION:
Main goal The aim is to further improve the inter-laboratory variability for the TGA-CAT (Thrombin generation assay-calibrated automated thrombogram) method by using an elaborate standardization protocol and in extension making the use of large prospective multi-center studies a reality.

Goals of the project are:

* To determine the inter-laboratory variability by evaluating an enhanced standardized TGA-CAT protocol.
* To evaluate if the inter-laboratory variability of the TGA-CAT method is effected by administration of a recombinant FVIII product (Advate) in a person with severe hemophilia A
* To evaluate if the inter-laboratory variability of the TGA-CAT method is effected by administration of a long acting FVIII product (Adynovate) in a person with severe hemophilia A
* To evaluate three reference plasma´s ability, through normalization of data, to improve the lab-to-lab variability.

Introduction The TGA CAT method has proved its usefulness for multiple purposes including diagnosis and management of bleeding disorders (1, 2), detecting hyper coagulability (3, 4), and monitoring and characterization of oral anticoagulant drugs (5, 6). Most of these studies are single-center studies and large prospective multi-center studies are needed to further validate the results. These multi-center studies have proved to be hard to produce due to lack of standardization of the method. In the last couple of years several articles have addressed the problem with large inter-laboratory variability for the TGA-CAT method by presenting thoroughly worked-out standardization protocols. Focus has been put both on the method itself and its pre-analytical factors as well as the usage of reference plasmas (RP) for normalization of results. One article showed that the choice of RP for the normalization of results could greatly reduce the inter-lab variability and that certain RP have a better ability to do so (7).

Lately a number of recombinant Factor VIII (rFVIII) and IX (rFIX) drugs with prolonged half-life have been developed and are about to or even have reached the market. The length of the pro-longed activity of the drug differs between patients and a need for individual tailoring of the patient´s drug administration is obvious. Thrombin generation could prove to be an excellent tool in tailoring the optimal drug administration and monitoring the effect of the drug for each individual.

Methods and materials Thrombin generation Thrombin generation will be measured according to the method described by Hemker et al.(8): calibrated automated thrombogram (CAT, Thrombinoscope BV, Maastricht, the Netherlands).

Reagents PPP-reagent LOW (1 pM), PPP-reagent (5 pM), Thrombin Calibrator and FluCa-kit (TS31.00, TS30.00, TS20.00 and TS50.00, Thrombinoscope BV, Maastricht, The Netherlands) will be used in the test.

Samples Three different plasmas will be tested, normal plasma, hypo- and hypercoagulable plasma. Normal and hypercoagulable plasma will be pooled from 3 donors and hypocoagulable plasma will be collected from 4 donors. Hypocoagulable plasma will be collected from five haemophilia A (HA) patients regularly treated at the Malmö Coagulation Unit by taking 10 4.5 mL tubes of citrated blood at one occasion. Normal plasma will be collected from 3 co-workers at the same unit, each person donating 13 tubes of 4.5 mL citrated blood. Hypercoaguable plasma will be prepared from 3 healthy volunteers, shown to have TGA CAT parameter values >2 SD of median by taking 13 tubes of 4.5 mL citrated blood. Plasma from one patient with severe HA patient that have been given FVIII-concentrates, Advate™ respectively the long-acting Adynovate™ at two separate occasions will also be tested. After informed consent the patient will be asked not to take his regular profylaxis dose for 72 hours. The patient will be given Advate™ and Adynovate™ respectively at 30 U/kg. The monitoring samples will be taken 1h, 8h, 24h, 36h and 48h (Advate™) and 1h, 24h, 36h, 48h and 72h (Adynovate™) after injection. At each time point 3 tubes of 4.5 mL blood will be taken.

Reference plasmas Siemens Control Plasma P diluted 1:5 will be used as hypocoaguable RP, HemosIL calibration plasma (Instrumentation Laboratory, Bedford, Ma, USA) will be used as Standard RP and as hypercoagable plasma PS-DP (protein S-deficiency plasma)(Enzyme research laboratories, South Bend, In, USA) will be used.

Statistical analysis Raw data will be collected and analyzed at the Coagulation Unit, Skåne University Hospital, Malmö. Each participating center will be matched with Malmö Coagulation unit in a test of agreement where Bland-Altman bias plot will be used. The mean, standard deviation (SD) and coefficient of variation (CV%) will be calculated for each center with and without normalization and displayed in a table. The Advate/ Adynovate elimination profiles will be plotted and multivariate repeated measurements analyses of variance including a general test for parallel curves, will be applied to evaluate differences between Centers in the elimination profiles.

Study design The study aims to evaluate the inter-laboratory variability of TGA-CAT performed TGT with a highly standardized protocol, how the use of RFs for normalization of data impact on variability of results and to evaluate the usefulness of TGA-CAT in monitoring prolonged FVIII drug administration. All Fluorometers of the participating center´s should be serviced and have temperature calibrated to 37 C prior start of the study. The latest software version must be installed (Thromboscope BV, Maastricht, The Netherlands, version V5.0.0.742). All laboratory equipment, pipettes, water baths, water purifiers, etc., needs to be calibrated. All plasmas, TGA-CAT reagents needed for the study will be administered and distributed to all participating centers by the Coagulation Unit, Malmö. An USB-memory stick containing a plate set-up scheme file and a video file covering critical pre-analytical and analytical steps will also be provided alongside the samples and reagents. Three pooled plasmas (normal, hypo- and hypercoaguable), three RF, five Adynovate and five Advate monitoring samples will be run five times on five different days by each participating center, following a scheme provided in the USB-memory stick, with two different triggers, PPP-reagent LOW (1 pM) and PPP-reagent (5 pM). Two test runs are scheduled each day to maximize RF and reagent usage. The reason for testing three different types of RF is the fact an earlier study results implied a better reduction of variability when using, for an example a hypocoaguable RF to hypocoaguable plasmas (9).

ELIGIBILITY:
Inclusion Criteria:

* For patients with severe hemophilia A (study group 1)(n=4) that has not received any factor concentrate within 72 hours: Diagnosis of severe hemophilia, with regular check-ups at the hemophilia center at SUS, Malmö and willingness to participate
* For healthy controls (n=3) (study group 2): Willingness to participate
* For healthy controls with a documented high TGC (study group 3): Willingness to participate

Exclusion Criteria

* For patients with severe hemophilia A (study group 1)(n=4) that has not received any factor concentrate within 72 hours: Intake of any other pharmaceutical product known to have an effect on the coagulation system the last 14 days, to the judgement of the including investigator
* For healthy controls (n=3) (study group 2): Any disorder known to affect the coagulation system and intake of any drug known to affect the coagulation system the last 14 days before blood sampling , to the judgement of the including investigator.
* For healthy controls with a documented high TGC (study group 3): Any disorder known to affect the coagulation system and intake of any drug known to affect the coagulation system within the last 14 days before blood sampling, to the judgement of the including investigator.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Patient with severe hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Inter lab variability | May 2017
  Coefficient of Variation (CV) i plasma samples with high, normal and low thrombin genration capacity
Inter lab variability | May 2017
  Coefficient of Variation (CV) i plasma samples from a patient treated with Advate
Inter lab variability | May 2017
  Coefficient of Variation (CV) and level of agreement i plasma samples from a patient treated with Adynovate

SECONDARY OUTCOMES:
Inter lab variability | May 2017
  Coefficient of Variation (CV) and level of agreement when results have been noramlized with plasma with high, normal and low thrombin generation capacity

CONTACTS AND LOCATIONS:
Overall Officials: Jan Astermark, MD PhD, Study Director — Department of hematology, Skane University hospital
Locations (1):
- Coagulation Unit, department of translational medicine, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Nair SC, Dargaud Y, Chitlur M, Srivastava A. Tests of global haemostasis and their applications in bleeding disorders. Haemophilia. 2010 Jul;16 Suppl 5:85-92. doi: 10.1111/j.1365-2516.2010.02304.x. PMID 20590862
- [Background] Trossaert M, Regnault V, Sigaud M, Boisseau P, Fressinaud E, Lecompte T. Mild hemophilia A with factor VIII assay discrepancy: using thrombin generation assay to assess the bleeding phenotype. J Thromb Haemost. 2008 Mar;6(3):486-93. doi: 10.1111/j.1538-7836.2007.02861.x. Epub 2007 Nov 28. PMID 18047548
- [Background] Dargaud Y, Trzeciak MC, Bordet JC, Ninet J, Negrier C. Use of calibrated automated thrombinography +/- thrombomodulin to recognise the prothrombotic phenotype. Thromb Haemost. 2006 Nov;96(5):562-7. PMID 17080211
- [Background] Lecompte T, Wahl D, Perret-Guillaume C, Hemker HC, Lacolley P, Regnault V. Hypercoagulability resulting from opposite effects of lupus anticoagulants is associated strongly with thrombotic risk. Haematologica. 2007 May;92(5):714-5. doi: 10.3324/haematol.10577. PMID 17488705
- [Background] Freyburger G, Macouillard G, Labrouche S, Sztark F. Coagulation parameters in patients receiving dabigatran etexilate or rivaroxaban: two observational studies in patients undergoing total hip or total knee replacement. Thromb Res. 2011 May;127(5):457-65. doi: 10.1016/j.thromres.2011.01.001. Epub 2011 Jan 31. PMID 21277622
- [Background] Hacquard M, Perrin J, Lelievre N, Vigneron C, Lecompte T. Inter-individual variability of effect of 7 low molecular weight antithrombin-dependent anticoagulants studied in vitro with calibrated automated thrombography. Thromb Res. 2011 Jan;127(1):29-34. doi: 10.1016/j.thromres.2010.07.024. Epub 2010 Sep 17. PMID 20850172
- [Background] Dargaud Y, Luddington R, Gray E, Lecompte T, Siegemund T, Baglin T, Hogwood J, Regnault V, Siegemund A, Negrier C. Standardisation of thrombin generation test--which reference plasma for TGT? An international multicentre study. Thromb Res. 2010 Apr;125(4):353-6. doi: 10.1016/j.thromres.2009.11.012. Epub 2009 Nov 26. PMID 19942257
- [Background] Perrin J, Depasse F, Lecompte T; French-speaking CAT group and under the aegis of GEHT; French-speaking CAT group (all in France unless otherwise stated):; French-speaking CAT group all in France unless otherwise stated. Large external quality assessment survey on thrombin generation with CAT: further evidence for the usefulness of normalisation with an external reference plasma. Thromb Res. 2015 Jul;136(1):125-30. doi: 10.1016/j.thromres.2014.12.015. Epub 2014 Dec 24. PMID 25563679
- [Background] Hemker HC, Giesen P, Al Dieri R, Regnault V, de Smedt E, Wagenvoord R, Lecompte T, Beguin S. Calibrated automated thrombin generation measurement in clotting plasma. Pathophysiol Haemost Thromb. 2003;33(1):4-15. doi: 10.1159/000071636. PMID 12853707